CLINICAL TRIAL: NCT05421416
Title: Loratadine for the Prevention of Bone Pain Caused by Granulocyte Colony Stimulating Factor (G-CSF) During Stem Cell Mobilization
Brief Title: Loratadine for the Prevention of G-CSF-related Bone Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IIT-0020
Record Dates: First submitted 2022-06-10; First posted 2022-06-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Stem Cell Transplant Complications
MeSH Terms: interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Loratadine Arm (Experimental): Loratadine 10mg, administered initially 3 hours before the first dose of G-CSF in the autologous stem cell mobilization protocol, and then daily for a minimum of 8 days.
  Interventions: Drug: Loratadine
- Placebo Arm (Placebo Comparator): Placebo capsule, administered initially 3 hours before the first dose of G-CSF in the autologous stem cell mobilization protocol, and then daily for a minimum of 8 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Loratadine — Loratadine is 2nd generation inverse agonist that exerts its effect by targeting H1 histamine receptors.
  Arms: Loratadine Arm
Drug: Placebo — Placebo sugar pill
  Arms: Placebo Arm

SUMMARY:
The research question for the current study is: Is loratadine more effective than placebo in preventing G-CSF-related bone pain during autologous hematopoetic stem cell transplant in patients with lymphoma or multiple myeloma? The hypothesis is that prophylaxis with loratadine will help prevent or reduce the severity of bone pain in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. A histologically or cytologically documented lymphoma or multiple myeloma
2. Next line of therapy is autologous stem cell transplant
3. Adult ≥ 18 years old.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
5. Life expectancy of at least 12 weeks.
6. The absence of any additional poorly controlled systemic disease that is directly contraindicated or places subject at significant risk, including but not limited to: congestive heart failure, diabetes mellitus, cirrhosis or liver failure, renal failure.
7. Able to adhere to study protocols and visit schedules

Exclusion Criteria:

1. Hypersensitivity or intolerance to antihistamines
2. Use of antihistamines within two days prior to the study period, excepting the use of single dose antihistamines during chemotherapy or blood transfusion protocols.
3. Recent use of G-CSF or pegfilgrastim defined as within 12 weeks of study accrual.
4. New and continued regular use of analgesics within the four days prior to the first dose of G-CSF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Bone Pain Severity (Brief Pain Inventory) | Brief Pain Inventory will be completed at baseline, daily during treatment (up to 12 days) and at the end of treatment (max day 12).
  Reduction in bone pain will be measured as a change from pre-G-CSF baseline in the Brief Pain Inventory (BPI), with median values compared for each trial arm. BPI pain severity will be compared as a composite score (sum of individual pain values divided by 4).
Bone Pain Interference (Brief Pain Inventory) | Brief Pain Inventory will be completed at baseline, daily during treatment (up to 12 days) and at the end of treatment (max day 12).
  Reduction on impact on daily life as a composite score out of 10 as measured on the Brief Pain Inventory (BPI). BPI pain interference will be compared as a composite score (sum of individual pain interference values divided by 7).
Bone pain severity (QLQ-BM22) | QLQ-BM22 will be completed at baseline and at the end of treatment (max day 12).
  Change in bone pain measured pre and post G-CSF in EORTC QLQ-BM22. QLQ-BM22 questionnaires will be compared to the post vs pre-treatment values and calculated as a composite sum (i.e. pre-treatment total score subtracted from post-treatment total score).

SECONDARY OUTCOMES:
Stem cell mobilization efficacy | Single measurement at the end of mobilization protocol (max day 8)
  Normalized mean and absolute number number of stem cells collected at the end of the mobilization protocol
Mean time to stem cell re-engraftment | Single measurement during stem cell re-infusion (max day 8)
  Time in days between stem cell re-infusion and the measurement on complete blood count (CBC) of an absolute neutrophil count of greater than 500/mm3 for 3 consecutive days.
Rate of plerixafor use during in each study arm | Single measurement after all patients have completed end of treatment.
  Proportion of patients in each study arm that require use of plerixafor during stem cell mobilization
Rate of pain control use | Single measurement after all patients complete mobilization (max day 8)
  Proportion of patients in each study arm that require use of additional pain control methods while receiving G-CSF.
Qualitative breakthrough of pain control use | Qualitative description of analgesic type after all patients complete mobilization (max day 8)
  Type of medication used to control additional pain while receiving G-CSF.
Progression free survival | Patients will be followed for 1 year after completion of the study treatment.
  Time between the date of treatment initiation and the date of disease progression or death (whatever the cause), whichever occurs first)

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided